CLINICAL TRIAL: NCT05890092
Title: Vulvar Disease in Nigeria - Registry ( Observationsl Study)
Brief Title: Vulvar Disease in Nigeria Observational Study
Acronym: VdiN
Status: Recruiting | Type: Observational
Sponsor: KDRS ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: KDRS-NGR001
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Vulvar Diseases; Vulvar Atrophy; Dermatoses
MeSH Terms: conditions — Vulvar Diseases; Skin Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — Observing for disease prevalence - actual and self-reported

SUMMARY:
Vulvar disease in Nigeria A look at awareness within patients and health practitioners, self-reported and actual prevalence within communities in Nigeria

ELIGIBILITY:
Inclusion Criteria:

* biological females - afab

Exclusion Criteria:

* none-afab

Ages: 10 Years to 90 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: All afab, willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Vulvar disease | 1-12 months
  Awareness of Vulvar disease (descriptor)

CONTACTS AND LOCATIONS:
Locations (1):
- Kdrs, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided